CLINICAL TRIAL: NCT05851508
Title: A Multicenter, Double-blinded, Randomized, Placebo-controlled Trial to Compare the Effectiveness of Intratympanic Injections methylPREDnisolon Versus Placebo in the Treatment of Vertigo Attacks in MENière's Disease (PREDMEN Trial).
Brief Title: The Effecttiveness of Intratympanic Methylprednisolon Injections Compared to Placebo in the Treatment of Vertigo Attacks in Meniere's Disease
Acronym: PREDMEN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Gelre Hospitals (Other); Maasstad Hospital (Other); Maastricht University Medical Center (Other); Medisch Spectrum Twente (Other); HagaZiekenhuis (Other)
Responsible Party: Principal Investigator, Babette F van Esch, MD, PhD, dr. van Esch, MD, PHD, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PREDMEN; 10140022110009 (Other Grant/Funding Number: ZonMW)
Record Dates: First submitted 2023-02-20; First posted 2023-05-09 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Meniere Disease
Keywords: Meniere's disease; Methylprednisolon; Intratimpanic corticosteroids; Dizziness; Hearing loss; tinnitus; aural fullness; randomized control trial
MeSH Terms: conditions — Meniere Disease; Dizziness; Hearing Loss; Tinnitus | interventions — Methylprednisolone

STUDY DESIGN:
Intervention Model Description: A multicenter, double-blinded, randomized, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Trial subjects, treating physicians and outcome assessors will be blinded throughout the entire study. Pharmacy staff will be unblinded for randomization and treatment allocation.
  Emergency unblinding may occur in the following situations: in case of a medical emergency where knowledge of the blinded treatment is necessary, for the treatment of (serious) adverse event, in the event of a SUSAR (Suspected Unexpected Serious Adverse Reaction) needing expedited reporting or if requested by the Safety Committee.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methylprednisolon (Active Comparator): Intratympanal injection with Methylprednisolon 62.5 mg/ ml
  Interventions: Drug: Methylprednisolon
- Placebo (Placebo Comparator): Intratympanal injection with saline, natriumchloride 0.9%
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylprednisolon — Intratympanal injection with Methylprednisolon 62.5 mg/ ml
  Arms: Methylprednisolon
Drug: Placebo — Intratympanal injection with saline, natriumchloride 0.9%
  Arms: Placebo

SUMMARY:
Ménière's disease is an inner ear disorder in which patients suffer from attacks of vertigo, tinnitus and hearing loss. To date, it is unclear what the best treatment for this condition is. Giving injections in the inner ear with the adrenal cortical hormone methylprednisolone is a treatment that is already widely used, but still there is insufficient evidence in the effectiveness of this treatment. This multicenter trial compares a patient group which receives injections of methylprednisolone to a patient group which receives placebo injections. Subsequently, dizziness, tinnitus, hearing loss and quality of life will be assed and compared for the above mentioned groups, over a period of one year.

DETAILED DESCRIPTION:
Meniere's disease is an inner ear disease characterized by recurrent episodes of vertigo, hearing loss, tinnitus and aural fullness. It is estimated that 15000 patients in de Netherlands suffer from this disease. Endolymfactic hydrops is thought to be the underlying pathophysiology of the symptoms. Salt restriction, oral medication (diuretics and betahistine), intratympanic gentamicin and steroids, ablative surgery, and endolymphatic sac surgery are some of the current therapy options. A probable effectiveness of the treatment with intratympanic gentamicin is found but this treatment is ototoxic and carries a risk of hearing loss. Methylprednisolone injections have been shown to be safer, however there is insufficient data to support the efficacy of this treatment. Therefore in this double-blinded, randomized, placebo-controlled trial, effectiveness of intratympanic injections with methylPREDnisolon versus placebo in the treatment of vertigo attacks in MENière's disease is compared.

The investigators aim to include 74 patients in each arm, based on a statistical power of 80 percent. Patients will be randomly randomized to one of the two treatment arms, receiving either a placebo injection or a methylprednisolone sodium succinate injection at a dose of 62.5 mg/ml. After 14 days, this injection will be given once more. A follow-up visit will be scheduled after six and twelve months and telephone follow-up calls will be scheduled after three and nine months. The primary objective will be the control of vertigo, with secondary outcomes including hearing loss, tinnitus, the frequency of escape interventions, quality of life, adverse events and cost effectiveness.

ELIGIBILITY:
Inclusion criteria:

• Unilateral, definite MD according to the diagnostic criteria derived from the American Academy Otolaryngology Head and Neck Surgery, Classification Committee of the Bárány Society, European Academy of Otology and Neurotology and International Classification of Vestibular Disorders published in 2015 [7] (see Appendix 1):

Definite MD Two or more spontaneous episodes of vertigo, each lasting 20 minutes to 12 hours, AND Audiometrically documented low- to medium-frequency sensorineural hearing loss in one ear, defining the affected ear on at least one occasion before, during or after one of the episodes of vertigo, AND Fluctuating aural symptoms (hearing, tinnitus, or fullness) in affected ear (not better accounted for by another vestibular diagnosis)

* age > 18 years at the start of the trial.
* ≥ 4 vertigo attacks over the last 6 months.
* willing to adhere to daily trial medications and the follow-up assessments.

Exclusion criteria

A potential subject who meets any of the following criteria will be excluded:

* bilateral MD
* severe disability (e.g. neurological, orthopaedic, cardiovascular) or serious concurrent illness that might interfere with treatment or follow-up.
* active additional neuro-otologic disorders that may mimic MD (e.g. vestibular migraine, recurrent vestibulopathy, phobic postural vertigo, vertebro-basilar TIAs, acoustic neuroma).
* otitis media with effusion based on tympanogram results.
* history of intratympanic injections with corticosteroid less than 6 months ago.
* history of intratympanic injections with gentamicin or ear surgery for treating MD.
* pregnant women and nursing women.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Vertigo spells | Daily, change from baseline to one year
  A definitive vertigo spell is defined as a spontaneous rotational vertigo symptom, which lasts at least 20 minutes and is often accompanied by disequilibrium and vomiting. No loss of consciousness is present. Vertigo spells are measured daily with the dizzy quest ap. Futhermore, at baseline after 6 and 12 months, caloric testing and a video-head impusle test are performend. Additionally the dizziness handicap inventory will be taken.

SECONDARY OUTCOMES:
Hearing loss | At baseline, 6 months and 12 months
  Hearing loss will be measured at baseline, 6 and 12 months after injection. Pure tone audimetry and extended fletcher index including the speech discrimination score will be tested.
Tinnitus | At baseline, 6 months and 12 months
  Tinnitus will be measured with the tinnitus handicap inventory at baseline, after 6 and 12 months.
health-related quality of life | At baseline, 6 months and 12 months
  The health realted quality of life will be evaluated with the generic quality of life questionnaire: EQ-5D
health-related quality of life | At baseline, 6 months and 12 months
  The health realted quality of life will be evaluated with the generic quality of life questionnaire: EQ-VAS, this will be a scale from 0 to 100 in which 0 means the worst health you can imagine and 100 means the best health you can imagine
Escape medication | At baseline, 3 months, 6 months, 9 months, 12 months
  The frequency of use of metoclopramide in the acute phase of vertigo will be registered.
Adverse events | Daily, change from baseline to one year
  At each study visit, subjects will be questioned about adverse events they have experienced since the last study visit.
Cost-effectiveness | At baseline, 6 months and 12 months
  Costs per QALY, this will be calculated from above mentioned outcomes on quality of life.
Co-interventions | Daily, change from baseline to one year
  The use of additional methylprednisolon or gentamicine will be evaluated during the entire study.
Overall function | At baseline, 6 months and 12 months
  The functional level scale will be measured with the questionnaire: Functional level scale: a scale from 1-6 in which 1 means: my dizziness has no effect on my activities and 6 means: I have been disabled for one year or longer and/or I received compensation (money) because of y dizziness or balance problem.
Impact of Dizziness | Change from baseline to 6 months to 12 months
  The impact of dizziness will be measured with the questionnaire: Dizziness handicap inventory
Tinnitus severity | At baseline, 6 months and 12 months
  The tinnitus severety will be measured with the questionnaire: Tinnitus functional index

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Centre, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data after deidentification will be shared upon reasonable request with researchers who provide a methodologically sound proposal. For analyses to achieve aims as described in the approved proposal.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data will be accessible after publication of the data
Access Criteria: Data can be shared upon reasonable request for multiple purposes. Proposals should be directed to M.M.E.Boreel@lumc.nl. To share data we will use the data transfer agreement in line with the template provided by the LUMC

REFERENCES:
- [Derived] Boreel MME, van Esch B, Schermer TR, Mol BM, van Benthem PP, Bruintjes TD. The effectiveness of intratympanic injections with methylPREDnisolon versus placebo in the treatment of vertigo attacks in MENiere's disease (PREDMEN trial): a study protocol for a phase-3 multicentre, double-blinded, randomised, placebo-controlled trial. BMJ Open. 2024 Aug 29;14(8):e076872. doi: 10.1136/bmjopen-2023-076872. PMID 39209781